CLINICAL TRIAL: NCT05154032
Title: Examining the Differential Effects of Traditional Float-REST on Sleep and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2104298113
Record Dates: First submitted 2021-09-24; First posted 2021-12-10 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Sleep Quality
Keywords: Sleep; Sensory Deprivation Tank; Wearable Technology
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: All participants will complete the following design. Women who experience menstrual flow will be scheduled to ensure that flow occurs on weeks 4 and 8 for consistency.
  Baseline block (weeks 1-4): At intake, participants will complete up to 13 surveys, which includes two baseline questionnaires, & the first rendition of weekly and monthly surveys. Participants will complete daily surveys each morning & night, & wear wearable devices to monitor physiology during sleep. Additionally, a laboratory visit will occur once per week for completion of weekly surveys & cognitive assessments; monthly surveys will also be completed during the fourth week.
  Intervention block (weeks 5-8): Daily, weekly, & monthly activities described for the baseline block will continue. Additionally, during weeks 5-7, participants will complete three 60-minute Float-REST sessions per week; The final week of this block will only involve the daily, weekly & monthly activities plus an exit survey.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Traditional Float-REST Therapy (Experimental): Participants will utilize sensory deprivation tanks.
  Interventions: Other: Traditional Float-REST Therapy

INTERVENTIONS:
Other: Traditional Float-REST Therapy — Traditional Float-REST therapy uses sensory deprivation tanks that consist of a very large warm water enclosure with a high concentration of Epsom salt to create a completely buoyant environment. This, along with a combination of temperature that is kept equal to skin temperature (94 degrees), allows the participant to eliminate the gravitational effects on the body, and along with lack of sound and low to no light (depending on comfort) allows the brain and body to completely relax for augmented physical and mental recovery. The room will contain an intercom that allows participants to communicate with study personnel in the event they need assistance. Participants will undergo 60 minute sessions three times a week for 3 weeks.
  Other Names: Sensory Deprivation Tanks

SUMMARY:
The objective of this research study is to assess how the implementation of Float-REST affects sleep quality, sleep structure, nocturnal physiology, subjective wellness, recovery from stressors, and resultant effects on performance and well-being.

DETAILED DESCRIPTION:
Traditional flotation therapy (Float-REST; Flotation Restricted Environmental Stimulation Therapy) uses sensory deprivation tanks that consist of a very large warm water enclosure with a high concentration of Epsom salt to create a completely buoyant environment. This, along with a combination of temperature that is kept equal to skin temperature (94 degrees), allows the participant to eliminate the gravitational effects on the body, and along with lack of sound and low to no light (depending on comfort) allows the brain and body to completely relax for augmented physical and mental recovery. Previous studies have examined the effects of sensory-deprivation tanks on both subjective (e.g., perceived stress and anxiety, self-reported muscle soreness) and objective measures of recovery (e.g., blood pressure, skill performance) though findings are incomplete and contradictory. Additionally, provided the growing understanding that sleep quality and quantity are at the forefront of ensuring optimal human performance states, compounded by the deleterious effects of high stress and anxiety on sleep, utilizing flotation therapy as a mechanism for enhancing sleep requires further investigation.

To identify whether Float-REST influences sleep and related behaviors, an eight week design will be executed that comprises an initial four weeks of baseline data collections followed by four weeks of intervention application and measure. Intervention will consist of three 60 minute Float-REST sessions per week, for the first three weeks of the intervention block (weeks 5-7 of the study). Data measures include wearable device monitoring, surveys, and brief cognitive tasks that are collected at various timepoints throughout the study (intake, monthly, weekly, daily, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-50 years of age

Exclusion Criteria:

* Has undergone travel across more than two collective time zones in the last two weeks
* Has a head diameter outside the range of 20.8-24 inches, or an approved head-mounted EEG device doesn't otherwise fit properly
* Has undergone a float-REST session of any kind in the last 3 months
* Has a fresh piercings that is less than 6 weeks old from scheduled session
* Has a fresh tattoo that is less than 4 weeks old from scheduled float
* Has an injury requiring an orthopedic cast (i.e. plaster or synthetic), irremovable splint or brace
* Is claustrophobic (fear of confined spaces)
* Has a skin or respiratory sensitivity or allergy to chlorine, sulfate, and/or magnesium
* Has a history of or is prone to motion sickness
* Has had an episode of loss of consciousness in the last 6-months
* Has had a concussion or traumatic brain injury in the last 6-months
* Has a contagious skin condition Has skin ulcers, open rashes, incisions, stiches or large open wounds that could cause pain when exposed to saltwater
* Has an irremovable medical port or catheter
* Has had a seizure in the last 10 years
* Has communicable diseases (e.g. HIV, Hepatitis A, B & C, tuberculosis, or measles)
* Lack of control of bodily functions prior to scheduled float
* Is pregnant or actively trying to become pregnant
* Has a known or diagnosed sleep disorder
* Females who have become menopausal or are exhibiting signs or symptoms of becoming perimenopausal
* Females who are unable to identify when their monthly menstrual period will occur
* Individuals who work during the night shift or have significantly abnormal sleep schedule
* Individuals who intend to have any significant medical procedures scheduled to occur within 12 weeks of enrollment
* Individuals who have intentions, or have discussed with their doctor, about adding or making any alterations to their prescribed medications within 12 weeks of enrollment
* Individuals who have any travel plans or other obligations within 12 weeks of enrollment that would prevent them from completing study requirements and attending required laboratory visits
* Individuals who intend to make significant alterations to their sleeping patterns within 12 weeks of enrollment. This may include, but is not limited to, changes such as moving, getting a new mattress, having someone move in with them, etc.
* Does not meet the ACSM's guidelines for exercise prescription. This is defined as:

  1. Presenting with an absolute contraindication OR

     1. Has a known cardiovascular, pulmonary, renal, metabolic disease, or other chronic illness
     2. Presents with symptoms indicating cardiovascular, pulmonary, renal, or metabolic disease
  2. presenting with two or more relative contraindications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Change in Nocturnal Heart Rate as measured by OURA Ring | Daily from baseline through study completion at 8 weeks
  Heart rate (beats per minute) will be quantified throughout the night via the OURA ring.
Change in Sleep Quantity as measured by Electroencephalography | Daily from baseline through study completion at 8 weeks
  Sleep stage duration (and the cumulative sleep duration) will be quantified each night via the Dreem headband, which uses Electroencephalography (EEG) for automatic sleep stage scoring.
Change in Subjective Sleep Quality | Daily from baseline through study completion at 8 weeks
  A custom daily morning questionnaire will be used to record how a participant feels the quality of their sleep was the previous night (e.g. 1, very poor; 10 excellent). This questionnaire will be taken on the participants smartphone within 30 minutes of waking.
Change in Nocturnal Heart Rate Variability as measured by OURA Ring | Daily from baseline through study completion at 8 weeks
  Heart rate variability will be quantified throughout the night via the OURA ring.
Change in Anxiety surrounding Float-REST as measured by the State Trait Anxiety Index | Before and after each float session (Weeks 5-7)
  Participants will complete the previously validated State Trait Anxiety Index (STAI) before and after each float session as a measure of subjective anxiety, where higher scores are suggestive of greater anxiety.
  State-Trait Anxiety Index (STAI) - Commonly used measure of state and trait anxiety, and done with 20 very brief questions. Values range from 20 to 80, with higher scores representing more severe anxiety. Participants will complete the STAI questionnaire before and after each session. The sessions will take place during weeks 5-7.
Change in heart rate during Float-REST as measured via Electrocardiography | During each float session (weeks 5-7)
  Participants will be monitored throughout float sessions using a heart rate monitor that will capture trends in cardiovascular physiology throughout the session.
Change in heart rate variability during Float-REST as measured via Electrocardiography | During each float session (weeks 5-7)
  Participants will be monitored throughout float sessions using a heart rate monitor that will capture trends in cardiovascular physiology throughout the session.

SECONDARY OUTCOMES:
Change in Subjective Athens Insomnia Scale measured via questionnaire | Weekly throughout study completion at 8 weeks
  Participants will complete previously validated questionnaires as often as once weekly throughout the study period (8 weeks).
  Athens Insomnia Scale (AIS) - eight-item questionnaire assessing sleep behaviors on a scale of 0 to 3. Higher scores = greater difficulty.
Change in Subjective Epworth Sleepiness Scale measured via questionnaire | Weekly throughout study completion at 8 weeks
  Participants will complete previously validated questionnaires as often as once weekly throughout the study period (8 weeks).
  Epworth Sleepiness Scale (ESS) - eight-item questionnaire assessing sleep behaviors on a scale of 0 to 3. Higher scores = increased average sleep propensity in daily life
Change in Subjective Insomnia Severity Index measured via questionnaire | Weekly throughout study completion at 8 weeks
  Participants will complete previously validated questionnaires as often as once weekly throughout the study period (8 weeks).
  Insomnia Severity Index (ISI) - seven-item questionnaire assessing sleep behaviors on a scale of 0 to 3. Higher scores = increased severity.
Change in Subjective Restorative Sleep Questionnaire | Weekly throughout study completion at 8 weeks
  Participants will complete previously validated questionnaires as often as once weekly throughout the study period (8 weeks).
  Restorative Sleep Questionnaire (RSQ) - nine-item questionnaire assessing sleep behaviors on a scale of 0 to 5. Higher scores = better sleep
Change in Subjective Patient Reported Outcomes Measurement Information System measured via questionnaire | Weekly throughout study completion at 8 weeks
  Participants will complete previously validated questionnaires as often as once weekly throughout the study period (8 weeks).
  Patient Reported Outcomes Measurement Information System (PROMIS) - seven item questionnaire assessing sleep behaviors on a scale of 0 to 5. Higher scores = healthier subject
Subjective Sleep Preferences | Once at the beginning of week 1
  At intake, a custom baseline questionnaire will be completed to record each participants sleep preferences and common behaviors. These sleep preferences will be used to identify if Float-REST tends to be more or less successful for certain individuals based upon predetermined qualities.
Subjective Success of Float-REST | Once at the end of week 8
  Following completion of the study, a custom questionnaire will record how successful the participant believes Float-REST was for improving their sleep and well-being. Participants will indicate how much they relate to a particular item on a scale of "Not at all" to "Very much so"
Changes in Conflict Management via Questionnaire | Monthly from baseline through study completion at 8 weeks
  Participants ability to manage conflict and the strategies in which they approach conflict will be assessed via the Conflict Management Questionnaire. This questionnaire scores the management of various situations based upon the participant responses (definitely true, true, tends to be true, tends not to be true, not true, definitely not true) and classifies the highest scoring response category as being the participant's preferred method of handing conflict. Scores of the response categories will be compared.
Changes in Emotional Regulation as measured via Emotional Regulation Questionnaire | Monthly from baseline through study completion at 8 weeks
  Participants' ability to regulate their emotions appropriately will be quantified via the previously validated Emotional Regulation Questionnaire (ERQ), in which participants will indicate how much they agree with each statement (1, strongly disagree; 7, strongly agree).
Changes in Perceived Stress as measured via Perceived Stress Scale | Weekly from baseline through study completion at 8 weeks
  Participants' perceived stress will be quantified via the previously validated Perceived Stress Scale (PSS), which asks participants to report on the frequency of various experiences (0, never; 4, very often) and final scoring suggests lower scores to be associated with lower levels of stress.
Changes in Subjective Sleep as measured via Pittsburgh Sleep Quality Index | Monthly from baseline through study completion at 8 weeks
  Participant's subjective reports of sleep quality will be quantified through the previously validated Pittsburgh Sleep Quality Index (PSQI). Questions are scored into multiple components to determine sleep difficulty in various areas, where higher scores are indicative of greater sleep difficulties; these scores will be compared across timepoints.
Changes in Subjective Anxiety as measured via the State Trait Anxiety Index | Monthly from baseline through study completion at 8 weeks
  Participants will complete the previously validated State Trait Anxiety Index (STAI) as a measure of subjective anxiety, where higher scores are suggestive of greater anxiety.
Changes in Sleep Disturbances as measured via the Sleep Disorders Questionnaire | Monthly from baseline through study completion at 8 weeks
  Participants will complete a 34 item checklist that has been previously used for screening of a potential sleep disorder; the more items that the participant feels applies to them, the higher the likelihood of the individual having a sleep disorder.
Change in Cognitive Performance via Stroop Task | Weekly from baseline through study completion at 8 weeks.
  Participants will complete the Stroop Task at intake and once weekly throughout the study on a computer. The task requires participants to respond to the presentation of a word by clicking the key associated with the ink color rather than the meaning of the word. Participants will be monitored for speed and accuracy of responses.
Change in Response Inhibition via SART 2 | Weekly from baseline through study completion at 8 weeks.
  Participants will complete the SART 2 task at intake and once weekly throughout the study on a computer. The task requires participants to respond, or refrain from responding, to the presentation of a number; a predetermined number is provided at the start of the task that participants are asked to refrain from responding to. Participants will be monitored for speed and accuracy of responses.
Change in Attentional Vigilance via Mackworth Clock Task | Weekly from baseline through study completion at 8 weeks.
  Participants will complete the Mackworth Clock task at intake and once weekly throughout the study on a computer. The task requires participants to watch the second hand of a clock across five minutes and respond as quickly as possible to skips in the clock's second hand by pressing a key. Participants will be monitored throughout the task for speed and accuracy of responses.
Change in Mental Rotation via Computer Task | Monthly from baseline through study completion at 8 weeks.
  Participants will complete the Mental Rotation task at intake and once monthly throughout the study on a computer. The task requires participants to respond as quickly as possible by select from two pictures that accurately depicts the same object that is presented in a different position in a third picture. 10 warm up trials will be completed followed by 10 test trials. Participants will be monitored throughout the task for speed and accuracy of responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Rockefeller Neuroscience Institute at West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided